CLINICAL TRIAL: NCT04681482
Title: Effectiveness and Safety of Oral Anticoagulants Among Obese Patients With Non-Valvular Atrial Fibrillation in the Veterans Affairs Population With Medicare
Brief Title: Effectiveness And Safety Of Oral Anticoagulants Among Obese Patients With Non-Valvular A-Fib In VA Patients With Medicare
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B0661162
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Results first posted 2021-12-06 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Atrial Fibrillation; Obesity; Anticoagulants
Keywords: Medicare; Veterans Affairs; Major Bleeding; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Obesity; Stroke | interventions — apixaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Apixaban Group: The cohort prescribed apixaban and diagnosed with Atrial Fibrillation
  Interventions: Drug: Apixaban
- Warfarin Group: patients prescribed warfarin only diagnosed with Atrial Fibrillation.

INTERVENTIONS:
Drug: Apixaban — Anticoagulant medication used to treat and prevent blood clots and to prevent stroke in people with nonvalvular atrial fibrillation.
  Other Names: Eliquis
  Groups: Apixaban Group

SUMMARY:
The overall objective of this analysis is to understand patient characteristics, the use of treatment, and clinical outcomes among obese (overweight) and severely obese patients with non-valvular atrial fibrillation (NVAF) who initiate therapy with OACs (oral anti-coagulants). The aim of this study is to compare all DOACs (direct oral anti-coagulants) to warfarin.

However, the primary analysis will be conducted among apixaban vs warfarin patients only. If sample size permits, we will also conduct other DOAC vs warfarin and DOAC vs DOAC analysis.

ELIGIBILITY:
Inclusion Criteria:

* Obese or severely obese.
* Initiated an OAC from July 1, 2013 - December 31, 2017; the first DOAC pharmacy claim date during the identification period will be designated as the index date. The first warfarin prescription date will be designated as the index date for patients without any DOAC claim.
* Individuals ≥18 years old as of the index date.
* Had 6 months continuous health plan enrollment with medical benefits (Parts A & B) for at least 6 months pre-index date (baseline period).
* At least 1 diagnosis of AF prior to or on index date, identified by any medical claim associated with an International Classification of Diseases, Ninth Revision, Clinical Modification (ICD-9-CM) code of 427.31 or International Classification of Diseases, Tenth Revision, Clinical Modification (ICD-10-CM) code of I480-I482, and I4891.
* Had body weight or BMI value reported within ±6 months of the index date.

Exclusion Criteria:

* Had medical claims indicating a diagnosis or procedure of rheumatic mitral valvular heart disease, heart valve replacement/transplant, venous thromboembolism, or transient AF 6 months prior to or on the index date.
* Had hip/knee replacement surgery within 6 weeks prior to or on the index date.
* Were pregnant during the study period.
* Had an OAC prescription during the 6 months pre-index date.
* Had follow-up time equal to 0 days.
* Had more than one OAC on the index date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese or severely obese AF patients in the CMS Medicare and Veterans' Health Affairs (VHA) databases who were newly prescribed OACs between January 1, 2013 and December 31, 2017.
Sampling Method: Non-Probability Sample
Enrollment: 107383 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2020-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B0661162

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a retrospective population-based registry study. Data for participants diagnosed with non-valvular atrial fibrillation (NVAF) and treated with either oral anticoagulants (OAC [Warfarin]) or direct oral anticoagulants (DOAC [Apixaban, Dabigatran and Rivaroxaban]) retrieved from the Veterans Affairs (VA) Population and Centre for Medicare and Medicare Services (CMS) database from January 2013 to December 2017.
Pre-assignment Details: In this study, inverse probability of treatment weighted (IPTW) method was used in analysis of outcome measures to balance participant's characteristics among reporting groups. Baseline for this study was 6 months prior to the index date. The index date was the date of first prescription for an OAC (Warfarin) or DOAC (Apixaban, Dabigatran, and Rivaroxaban) pharmacy claim during the identification period from July 1, 2013 -December 31, 2017.
Groups:
- Warfarin: Participants diagnosed with NVAF, who initiated warfarin on the index date, were included in this cohort and their data from July 2013 to December 2017, available in VA and CMS database observed retrospectively. Index date was defined as the date of the first warfarin prescription for participants without any DOAC claim.
- Apixaban: Participants diagnosed with NVAF, who initiated apixaban on the index date, were included in this cohort and their data from July 2013 to December 2017, available in VA and CMS database observed retrospectively. Index date was defined as the date of the first DOAC pharmacy claim date during the identification period (July 1, 2013-December 31, 2017).
- Dabigatran: Participants diagnosed with NVAF, who initiated dabigatran on the index date, were included in this cohort and their data from July 2013 to December 2017, available in VA and CMS database observed retrospectively. Index date was defined as the date of the first DOAC pharmacy claim date during the identification period (July 1, 2013-December 31, 2017).
- Rivaroxaban: Participants diagnosed with NVAF, who initiated rivaroxaban on the index date, were included in this cohort and their data from July 2013 to December 2017, available in VA and CMS database observed retrospectively. Index date was defined as the date of the first DOAC pharmacy claim date during the identification period (July 1, 2013-December 31, 2017).
Period: Overall Study
Arm/Group | Warfarin | Apixaban | Dabigatran | Rivaroxaban
Started | 35051 | 38756 | 12148 | 21428
Completed | 35051 | 38756 | 12148 | 21428
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included obese or morbidly obese atrial fibrillation (AF) participants in the CMS and VA databases with newly prescribed OACs or DOACs between January 1, 2013 and December 31, 2017.
Groups:
- Total: Total of all reporting groups
Arm/Group | Warfarin | Apixaban | Dabigatran | Rivaroxaban | Total
Number analyzed (Participants) | 35051 | 38756 | 12148 | 21428 | 107383
Age, Customized [Count of Participants; unit: Participants]
  18-54 years | 182 | 94 | 88 | 105 | 469
  55-64 years | 1380 | 833 | 580 | 827 | 3620
  65-74 years | 12410 | 13037 | 6873 | 10070 | 42390
  75-79 years | 5817 | 6504 | 1741 | 3472 | 17534
  >=80 years | 15262 | 18288 | 2866 | 6954 | 43370
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 456 | 576 | 139 | 299 | 1470
  Male | 34595 | 38180 | 12009 | 21129 | 105913
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2086 | 2024 | 621 | 1172 | 5903
  White | 32246 | 35847 | 11184 | 19732 | 99009
  More than one race | 529 | 654 | 220 | 343 | 1746
  Unknown or Not Reported | 190 | 231 | 123 | 181 | 725
Number of Participants From Different Regions of United States [Count of Participants; unit: Participants] — In this baseline measure, number of participants from different regions of the United States were reported. The United States was divided into 5 regions: northeast, midwest, south, west, and other/unknown.
  Participants
    Northeast | 7016 | 6821 | 1887 | 3718 | 19442
    Midwest | 10498 | 10046 | 3008 | 5858 | 29410
    South | 11809 | 15311 | 5080 | 8398 | 40598
    West | 5576 | 6392 | 2134 | 3361 | 17463
    Other/Unknown | 152 | 186 | 39 | 93 | 470
Number of Participants Classified According to OAC Index Year [Count of Participants; unit: Participants] — In this baseline measure, number of participants were classified according to the index year in which they received OAC. Index year was defined as the year (2013-2017) in which the treatment was initiated for the participants.
  Participants
    2013 | 5090 | 395 | 974 | 1135 | 7594
    2014 | 9024 | 2548 | 2462 | 3996 | 18030
    2015 | 7770 | 6792 | 2178 | 4370 | 21110
    2016 | 7289 | 12705 | 3336 | 5600 | 28930
    2017 | 5878 | 16316 | 3198 | 6327 | 31719
Dose of the Index DOAC [Count of Participants; unit: Participants] — In this baseline measure, number of participants received a standard dose (apixaban - 5 milligram [mg], dabigatran - 150 mg, and rivaroxaban - 20 mg); a lower dose (apixaban - 2.5 mg, dabigatran - 75 mg, and rivaroxaban - 15 mg/10 mg); and other dose (rivaroxaban - 10 mg, dabigatran - 110 mg) based on initial prescription of DOAC were reported. Population: No participant for reporting arm 'warfarin' had dose of DOAC at index date, hence, for this reporting group no data was collected and reported.
  Participants
    number analyzed (Participants) | 0 | 38756 | 12148 | 21428 | 72332
    Standard Dose (5 mg Apixaban, 150 mg Dabigatran, 20 mg Rivaroxaban) | 0 | 30494 | 11411 | 16108 | 58013
    Lower Dose (2.5 mg Apixaban, 75 mg Dabigatran, 15 mg Rivaroxaban) | 0 | 8262 | 726 | 4550 | 13538
    Other Dose (10 mg Rivaroxaban , 110 mg Dabigatran) | 0 | 0 | 11 | 770 | 781
Body Weight [Count of Participants; unit: Participants] — In this baseline measure, number of participants with body weight in kilogram (Kg) were reported within +/- 6 months from the index date.
  Participants
    <=60 Kg | 871 | 1009 | 149 | 359 | 2388
    61-99 Kg | 22449 | 25698 | 6924 | 13225 | 68296
    100-119 Kg | 7102 | 7830 | 3094 | 4776 | 22802
    >=120 Kg | 3714 | 3261 | 1614 | 2478 | 11067
    Missing | 915 | 958 | 367 | 590 | 2830
Body Mass Index (BMI) [Count of Participants; unit: Participants] — In this baseline measure, number of participants with BMI in kilogram per square meters (kg/m^2) ranged from less than (<) 18.5 kg/m^2 to greater than (>) 40 kg/m^2 were reported within +/- 6 months from index date.
  Participants
    <18.5 kg/m^2 | 285 | 296 | 47 | 121 | 749
    (18.5-24.9) kg/m^2 | 5921 | 6890 | 1586 | 3158 | 17555
    (25-29) kg/m^2 | 8803 | 10490 | 3041 | 5563 | 27897
    (30-39) kg/m^2 | 10293 | 11425 | 4357 | 6923 | 32998
    >40 kg/m^2 | 2176 | 1746 | 896 | 1294 | 6112
    Missing | 7573 | 7909 | 2221 | 4369 | 22072
International Normalized Ratio (INR) [Count of Participants; unit: Participants] — In this baseline measure, number of participants with or without INR were reported.
  Participants
    Yes | 15304 | 9133 | 3561 | 3977 | 31975
    No | 19747 | 29623 | 8587 | 17451 | 75408
CHADS2 Score [Count of Participants; unit: Participants] — In this baseline measure, CHADS2 score was assessed by combining score of 5 risk factors (congestive heart failure [CHF] history, hypertension history, age >=75 years, diabetes mellitus history and stroke symptoms previously). Score ranged from 0-6, where "0" indicates low risk and "6" indicates high risk, where higher scores indicated more risk.
  Participants
    0 | 1424 | 1506 | 944 | 1352 | 5226
    1 | 6829 | 7280 | 3640 | 5413 | 23162
    2 | 11372 | 12318 | 3985 | 6935 | 34610
    >=3 | 15426 | 17652 | 3579 | 7728 | 44385
CHA2DS2-VASc Score [Count of Participants; unit: Participants] — In this baseline measure, CHA2DS2-VASc score was assessed by combining score of 8 risk factors (CHF, hypertension, age >=75 years, diabetes mellitus, stroke [non-hemorrhagic only and transient ischemic attack {TIA}], vascular disease [myocardial infarction, peripheral arterial disease, aortic plaque], age 65 to 74 years, and sex category). Score ranged from 0-9, where "0" indicates low risk and "9" indicates high risk, where higher scores indicated more risk.
  Participants
    0 | 79 | 70 | 71 | 87 | 307
    1 | 1280 | 1405 | 886 | 1227 | 4798
    2 | 4703 | 5764 | 2709 | 4007 | 17183
    3 | 8196 | 9734 | 3520 | 5718 | 27168
    >=4 | 20793 | 21783 | 4962 | 10389 | 57927
HAS-BLED Score [Count of Participants; unit: Participants] — In this baseline measure, HAS-BLED score was assessed by combining score of 8 risk factors (hypertension, abnormal kidney or/liver function, age >=75 years, stroke, bleeding, labile INR, age >65 years, and alcohol/drug therapy). Score ranged from 0-9, where "0" indicates low risk and "9" indicates high risk, where higher scores indicated more risk.
  Participants
    0 | 135 | 109 | 83 | 130 | 457
    1 | 3859 | 4522 | 1733 | 2770 | 12884
    2 | 11444 | 13675 | 5457 | 8533 | 39109
    >=3 | 19613 | 20450 | 4875 | 9995 | 54933
Baseline Medication Use [Count of Participants; unit: Participants] — In this baseline measure, number of participants on medications prescribed at baseline were reported. Prescribed medications were angiotensin-converting enzyme (ACE) inhibitors/ angiotensin-receptor blockers (ARB), beta blockers, H2 receptor-antagonist, proton pump inhibitor, statins, anti-platelets, and non-steroidal anti inflammatory drugs (NSAIDS).
  Participants
    ACE/ARB | 13562 | 14295 | 4777 | 8049 | 40683
    Beta blockers | 18486 | 20198 | 6177 | 11211 | 56072
    H2-receptor antagonist | 2268 | 2584 | 695 | 1288 | 6835
    Proton pump inhibitor | 12227 | 13793 | 3896 | 7178 | 37094
    Statins | 23095 | 25830 | 7959 | 13901 | 70785
    Anti-platelets | 8686 | 10515 | 2980 | 5141 | 27322
    NSAIDS | 3819 | 5319 | 1904 | 3388 | 14430
Bariatric Surgery [Count of Participants; unit: Participants] — In this baseline measure, number of participants with bariatric surgery at baseline were reported.
  Participants | 130 | 125 | 43 | 93 | 391
Comorbid Conditions [Count of Participants; unit: Participants] — In this baseline measure, number of participants with various comorbid conditions such as bleeding history, CHF, diabetes mellitus, hypertension, renal disease, liver disease, myocardial infarction, dyspepsia or stomach discomfort, non-stroke/systemic embolism (SE) peripheral vascular disease, stroke/SE, TIA, anemia and coagulation defects, alcoholism, peripheral artery disease, and coronary artery disease were reported.
  Participants
    Bleeding History | 6021 | 5564 | 1367 | 2886 | 15838
    CHF | 13188 | 12385 | 3025 | 6062 | 34660
    Diabetes Mellitus | 15527 | 15225 | 4714 | 8453 | 43919
    Hypertension | 29689 | 32639 | 10117 | 17961 | 90406
    Renal Disease | 4540 | 8022 | 929 | 2367 | 15858
    Liver Disease | 1430 | 1388 | 418 | 814 | 4050
    Myocardial Infarction | 5344 | 5628 | 1200 | 2841 | 15013
    Dyspepsia or Stomach Discomfort | 4322 | 4201 | 1110 | 2438 | 12071
    Non-stroke/SE Peripheral Vascular Disease | 8994 | 9560 | 2276 | 4836 | 25666
    Stroke/SE | 4468 | 4731 | 1062 | 2186 | 12447
    TIA | 2750 | 4508 | 840 | 1807 | 9905
    Anemia and Coagulation Defects | 10572 | 9987 | 2129 | 4640 | 27328
    Alcoholism | 11323 | 14181 | 4241 | 7567 | 37312
    Peripheral Artery Disease | 8817 | 8927 | 2156 | 4610 | 24510
    Coronary Artery Disease | 19283 | 21041 | 5664 | 10903 | 56891

OUTCOME MEASURES:

1. Primary Outcome: Event Rate Per 100 Participant-Years For First Occurrence of Major Bleeding Events After Index Date in Obese Participants
Description: Event rate per 100 participant-years for first occurrence of major bleeding (MB) event after index date in obese participants was reported. MB after index date was identified using hospital claims and occurred anytime during the follow-up period of drug use or within 30 days from the last day of treatment prescription. Index date was defined as date of first DOAC pharmacy claim date during the identification period (July 1, 2013-December 31, 2017 [3.5 years]). The first warfarin prescription date was designated as the index date for participants without any DOAC claim. MB events included the composite of gastrointestinal (GI), intracranial hemorrhage (ICH), and other sites. MB was equal to 1 if bleeding event was greater than equal to (>=) 1.
Time Frame: From first dose of study drug to follow-up period or within 30 days from last prescription date (data collected and observed retrospectively for 3.5 years)
Population: Obese participants with or without DOAC treatment diagnosed with NVAF were included in the outcome measure. Analysis performed using IPTW method to balance participant characteristics among reporting groups.
Measure: Number; unit: Events Per 100 Participant-Years
Arm/Group | Warfarin | Apixaban
Number analyzed (Participants) | 12918 | 13604
Events Per 100 Participant-Years | 7.27 | 4.06
Statistical Analysis 1: Comparison: Warfarin vs Apixaban; Cox Proportional Hazards Model was used to compare the risk of MB between cohorts; Test type: Superiority; p < 0.001, Cox Proportional Hazards Model; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.54 to 0.70]

2. Primary Outcome: Event Rate Per 100 Participant-Years For First Occurrence of Major Bleeding Events After Index Date in Morbidly Obese Participants
Description: Event rate per 100 participant-years for first occurrence of MB event after index date in morbidly obese participants was reported. MB after index date was identified using hospital claims and occurred anytime during the follow-up period of drug use or within 30 days from the last day of treatment prescription. Index date was defined as date of first DOAC pharmacy claim date during the identification period (July 1, 2013-December 31, 2017). The first warfarin prescription date was designated as the index date for participants without any DOAC claim. MB events included the composite of GI, ICH, and other sites. MB was equal to 1 if bleeding event was >=1.
Time Frame: as for outcome 1
Population: Morbidly obese participants with or without DOAC treatment diagnosed with NVAF were included in the outcome measure. Analysis performed using IPTW method to balance participant characteristics among reporting groups.
Measure: Number; unit: Events Per 100 Participant-Years
Arm/Group | Warfarin | Apixaban
Number analyzed (Participants) | 2176 | 1746
Events Per 100 Participant-Years | 5.52 | 3.94

3. Primary Outcome: Event Rate Per 100 Participant-Years For First Occurrence of Stroke or Systemic Embolism (SE) Events After Index Date in Obese Participants
Description: Event rate per 100 participant-years for first occurrence of stroke or SE events after index date in obese participants was reported. Stroke/SE were identified using hospital claims and occurred anytime during the period of drug use or within 30 days from the last day of treatment prescription. Index date was defined as date of first DOAC pharmacy claim date during the identification period (July 1, 2013-December 31, 2017). The first warfarin prescription date was designated as the index date for participants without any DOAC claim. Stroke events included the composite of any ischemic, any hemorrhagic and SE stroke events. Stroke/SE was equal to 1 if stroke event was >=1.
Time Frame: as for outcome 1
Population: Obese participants with or without DOAC treatment diagnosed with NVAF were included in this outcome measure. Analysis performed using IPTW method to balance participant characteristics among reporting groups.
Measure: Number; unit: Events Per 100 Participant-Years
Arm/Group | Warfarin | Apixaban
Number analyzed (Participants) | 12918 | 13604
Events Per 100 Participant-Years | 2.09 | 1.51
Statistical Analysis 1: Comparison: Warfarin vs Apixaban; Cox Proportional Hazards Model was used to compare the risk of stroke/SE between cohorts; Test type: Superiority; p = 0.088, Cox Proportional Hazards Model; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.66 to 1.03]

4. Primary Outcome: Event Rate Per 100 Participant-Years For First Occurrence of Stroke or Systemic Embolism (SE) Events After Index Date in Morbidly Obese Participants
Description: Event rate per 100 participant-years for first occurrence of stroke or SE events after index date in morbidly obese participants was reported. Stroke/SE were identified using hospital claims and occurred anytime during the period of drug use or within 30 days from the last day of treatment prescription. Index date was defined as date of first DOAC pharmacy claim date during the identification period (July 1, 2013-December 31, 2017). The first warfarin prescription date was designated as the index date for participants without any DOAC claim. Stroke events included the composite of any ischemic, any hemorrhagic and SE stroke events. Stroke/SE was equal to 1 if stroke event was >=1.
Time Frame: as for outcome 1
Population: Morbidly obese participants with or without DOAC treatment diagnosed with NVAF were included in this outcome measure. Analysis performed using IPTW method to balance participant characteristics among reporting groups.
Measure: Number; unit: Events Per 100 Participant-Years
Arm/Group | Warfarin | Apixaban
Number analyzed (Participants) | 2176 | 1746
Events Per 100 Participant-Years | 1.51 | 0.92

5. Primary Outcome: Event Rate Per 100 Participant-Years For First Occurrence of Net Clinical Benefit After Index Date in Obese Participants
Description: Event rate per 100 participant-years for first occurrence of net clinical benefit after index date in obese participants was reported. For participants with stroke/SE or MB event, net clinical benefit was assessed by evaluating the first hospital claim for a stroke/SE or MB event. The hospital claim occurred anytime during the period of drug use or within 30 days from the last day of supply of treatment prescription. Index date was defined as date of first DOAC pharmacy claim date during the identification period (July 1, 2013-December 31, 2017). The first warfarin prescription date was designated as the index date for participants without any DOAC claim.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Number; unit: Event Rate Per 100 Participant-Years
Arm/Group | Warfarin | Apixaban
Number analyzed (Participants) | 12918 | 13604
Event Rate Per 100 Participant-Years | 8.44 | 5.12
Statistical Analysis 1: Comparison: Warfarin vs Apixaban; Cox Proportional Hazards Model was used to compare the risk of net clinical benefit between cohorts; Test type: Superiority; p < 0.001, Cox Proportional Hazards Model; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.60 to 0.76]

6. Primary Outcome: Event Rate Per 100 Participant-Years For First Occurrence of Net Clinical Benefit After Index Date in Morbidly Obese Participants
Description: Event rate per 100 participant-years for first occurrence of net clinical benefit after index date in morbidly obese participants was reported. For participants with stroke/SE or MB event, net clinical benefit was assessed by evaluating the first hospital claim for a stroke/SE or MB event. The hospital claim occurred anytime during the period of drug use or within 30 days from the last day of supply of treatment prescription. Index date was defined as date of first DOAC pharmacy claim date during the identification period (July 1, 2013-December 31, 2017). The first warfarin prescription date was designated as the index date for participants without any DOAC claim.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Number; unit: Event Rate Per 100 Participant-Years
Arm/Group | Warfarin | Apixaban
Number analyzed (Participants) | 2176 | 1746
Event Rate Per 100 Participant-Years | 6.48 | 4.52

7. Primary Outcome: Charlson Comorbidity Index (CCI)
Description: CCI based on various comorbid conditions such as myocardial infarction, CHF, peripheral vascular disease, cerebrovascular disease, dementia, chronic obstructive pulmonary disease, rheumatologic disease, peptic ulcer disease, mild liver disease, diabetes (mild to moderate), diabetes + complications, hemiplegia or paraplegia, renal disease, any malignancy (lymphoma and leukemia), moderate/severe liver disease, metastatic solid tumor, and acquired immune deficiency syndrome (AIDS) were reported. CCI score range was from 0 to 14, where "0"= low comorbid condition and "14"= high comorbid condition, higher scores indicated more comorbidity.
Time Frame: Baseline (6 months prior to index date)
Population: Analysis population included obese or morbidly obese AF participants in the CMS and VA databases with newly prescribed OACs or DOACs between January 1, 2013 and December 31, 2017.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Warfarin | Apixaban | Dabigatran | Rivaroxaban
Number analyzed (Participants) | 35051 | 38756 | 12148 | 21428
Units on a scale | 3.13 (2.68) | 2.55 (2.39) | 2.21 (2.18) | 2.49 (2.37)

8. Secondary Outcome: Time in Therapeutic Range (TTR) During Follow-up Period
Description: TTR was computed using INR values among warfarin participants during the follow-up. TTR was calculated based on the percentage of time a participant remained in therapeutic range evaluated during the entire follow-up period. TTR >=65 percent (%) was observed as good and TTR less than (<) 65% was observed as poor.
Time Frame: as for outcome 1
Population: TTR was calculated only for the warfarin arm, therefore data was not collected/observed for DOACs cohorts - apixaban, dabigatran, rivaroxaban.
Measure: Median (Full Range); unit: Percentage of time
Arm/Group | Warfarin
Number analyzed (Participants) | 35051
Percentage of time | 14 [0 to 1461]

ADVERSE EVENTS:
Description: Due to observational nature of study, minimum criteria for reporting adverse events did not met, hence adverse events were not collected
Arm/Group | Warfarin | Apixaban | Dabigatran | Rivaroxaban
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Data for Edoxaban drug cohort was not observed due to small sample size, based on Sponsor's decision. Data for creatinine clearance was not recorded and reported due to insufficient amount of data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/82/NCT04681482/Prot_SAP_000.pdf